CLINICAL TRIAL: NCT06528418
Title: Exploration and Study on the Identification of Various Pulmonary Diseases Using Volatile Organic Compounds Biomarkers in Human Exhaled Breath
Brief Title: Identification of Multiple Pulmonary Diseases Using Volatile Organic Compounds Biomarkers in Human Exhaled Breath
Status: Recruiting | Type: Observational
Sponsor: ChromX Health (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); First People's Hospital of Foshan (Other); Sichuan Cancer Hospital and Research Institute (Other); Liwan District Central Hospital (Unknown); Shanghai Chest Hospital (Other); Peking Union Medical College Hospital (Other); Guangzhou Development Zone Hospital (Unknown); Huangpu District Hongshan Street Community Health Service Center (Unknown); Huangpu District Chinese Medicine Hospital (Unknown); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Huangpu District Jiufo Street Community Health Service Center (Unknown); Huangpu District Xinlong Town Central Hospital (Unknown); Huangpu District Yonghe Street Community Health Service Center (Unknown); Huangpu District Lianhe Street Second Community Health Service Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: MLD001
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer; Lung Infection; COPD; Bronchitis; Pulmonary Fibrosis; Pulmonary Embolism; Pulmonary Arterial Hypertension; Pulmonary Tuberculosis; Pulmonary Abscess; Emphysema; Lung Injury; Cystic Fibrosis of the Lung; Bronchial Asthma; Bronchiectasis; Interstitial Lung Disease; Preserved Ratio Impaired Spirometry
Keywords: Pulmonary Disease; Volatile Organic Compounds; Human Exhaled Breath; micro Gas Chromatography-photoionisation; detector (μGC-PID) system
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Bronchitis; Pulmonary Fibrosis; Pulmonary Embolism; Pulmonary Arterial Hypertension; Tuberculosis, Pulmonary; Lung Abscess; Emphysema; Lung Injury; Cystic Fibrosis; Asthma; Bronchiectasis; Lung Diseases, Interstitial; Lung Diseases | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Volatile Organic Compounds in Human Exhaled Breath
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pulmonary disease: Individuals with abnormalities in lung CT imaging and clinically diagnosed with lung cancer, lung infection, chronic obstructive pulmonary disease (COPD), bronchitis, pulmonary fibrosis, pulmonary embolism, pulmonary arterial hypertension, tuberculosis, lung abscess, emphysema, radioactive lung injury, cystic fibrosis of the lung, Bronchial Asthma, Bronchiectasis, interstitial lung disease (ILD), preserved ratio impaired spirometry (PRISm) etc .
  Interventions: Other: Gas chromatography-mass spectrometry(GC-MS) and micro Gas Chromatography-photoionisation detector (μGC-PID) system
- normal individual: Individuals with no abnormalities detected in lung CT imaging.
  Interventions: Other: Gas chromatography-mass spectrometry(GC-MS) and micro Gas Chromatography-photoionisation detector (μGC-PID) system

INTERVENTIONS:
Other: Gas chromatography-mass spectrometry(GC-MS) and micro Gas Chromatography-photoionisation detector (μGC-PID) system — Exhaled breath samples from these participants will be collected and analyzed to detect volatile organic compound molecules in human exhaled breath by GC-MS and μGC-PID

SUMMARY:
The goal of this observational study is to develop an advanced expiratory algorithm model utilizing exhaled breath volatile organic compound (VOC) marker molecules. This model aims to accurately diagnose mutiple pulmonary diseases. The primary objectives it strives to accomplish are:

1. To assess the diagnostic accuracy of an exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model in diagnose several common pulmonary diseases.
2. To assess the diagnostic accuracy of an exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model in diagnose more pulmonary diseases.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional, observational cohort study aimed at recruiting 10,000 participants with multiple pulmonary disease, including lung cancer, lung infection, chronic obstructive pulmonary disease (COPD), bronchitis, pulmonary fibrosis, pulmonary embolism, pulmonary arterial hypertension, tuberculosis, lung abscess, emphysema, radioactive lung injury, cystic fibrosis of the lung, Bronchial Asthma, Bronchiectasis, interstitial lung disease (ILD), preserved ratio impaired spirometry (PRISm) etc . Exhaled breath samples from these participants will be collected and analyzed using Gas chromatography-mass spectrometry(GC-MS) and micro Gas Chromatography-photoionisation detector (μGC-PID) system. Upon obtaining the μGC-PID results, a comprehensive evaluation of the diagnostic capabilities of exhaled breath samples in differentiating various pulmonary diseases will be performed, leveraging clinical diagnostic results, CT examination data, and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age must be 18 years old or above.
* Patients must meet the CT imaging diagnostic criteria for different lung diseases, and patients must be able to provide electronic versions of CT image data.
* Patients must have a clear clinical diagnosis.
* All participants must sign a written informed consent form.

Exclusion Criteria:

* Pregnant women.
* Individuals with a history of cancer other than lung disease.
* Individuals who have undergone organ transplants or non-autologous (allogeneic) bone marrow or stem cell transplants.
* Individuals with other severe organic diseases or mental illnesses.
* Individuals with metabolic diseases such as diabetes, hyperlipidemia, etc.
* Any other condition that researchers deem unsuitable for participation in this clinical trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with abnormal lung CT images within the past six months, including lung cancer, lung infection, chronic obstructive pulmonary disease (COPD), bronchitis, pulmonary fibrosis, pulmonary embolism, pulmonary arterial hypertension, tuberculosis, lung abscess, emphysema, radioactive lung injury, cystic fibrosis of the lung, Bronchial Asthma, Bronchiectasis, interstitial lung disease (ILD), preserved ratio impaired spirometry (PRISm), etc .
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of an exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model in the diagnosis of several common pulmonary diseases. | 2 years
  The diagnostic performance of the exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model will be compared with clinical diagnosis and CT/LDCT diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

SECONDARY OUTCOMES:
The diagnostic accuracy of an exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model in the diagnosis of more pulmonary diseases. | 2 years
  The diagnostic performance of the exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model will be compared with clinical diagnosis and CT/LDCT diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

OTHER OUTCOMES:
Establish an exhaled breath VOC model for predicting specific gene mutations in some lung diseases. | 2 years
  Establish an exhaled breath VOC model for predicting specific gene mutations in some lung diseases. And evaluate the prediction accuracy by comparing the results of specific gene testing

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD Chronic Respiratory Disease Collaborators. Prevalence and attributable health burden of chronic respiratory diseases, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Respir Med. 2020 Jun;8(6):585-596. doi: 10.1016/S2213-2600(20)30105-3. PMID 32526187
- [Background] Ratiu IA, Ligor T, Bocos-Bintintan V, Mayhew CA, Buszewski B. Volatile Organic Compounds in Exhaled Breath as Fingerprints of Lung Cancer, Asthma and COPD. J Clin Med. 2020 Dec 24;10(1):32. doi: 10.3390/jcm10010032. PMID 33374433
- [Background] van de Kant KD, van der Sande LJ, Jobsis Q, van Schayck OC, Dompeling E. Clinical use of exhaled volatile organic compounds in pulmonary diseases: a systematic review. Respir Res. 2012 Dec 21;13(1):117. doi: 10.1186/1465-9921-13-117. PMID 23259710
- [Background] Wang J, Janson C, Gislason T, Gunnbjornsdottir M, Jogi R, Orru H, Norback D. Volatile organic compounds (VOC) in homes associated with asthma and lung function among adults in Northern Europe. Environ Pollut. 2023 Mar 15;321:121103. doi: 10.1016/j.envpol.2023.121103. Epub 2023 Jan 21. PMID 36690293
- [Background] V A B, Subramoniam M, Mathew L. Noninvasive detection of COPD and Lung Cancer through breath analysis using MOS Sensor array based e-nose. Expert Rev Mol Diagn. 2021 Nov;21(11):1223-1233. doi: 10.1080/14737159.2021.1971079. Epub 2021 Aug 27. PMID 34415806